CLINICAL TRIAL: NCT06825351
Title: A Feasibility Study of Psychological First Aid Versus Dialectal Behavioral Intervention in Undergraduate Students With Suicide Risk: A Comparative Crossover Randomized ControlledTrial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mahmoud Khedr, Dr Mahmoud Khedr, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025
Record Dates: First submitted 2025-02-09; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants: Undergraduate students identified as at risk for suicide. Interventions: Participants will receive both PFA and DBT at different times. PFA: Focuses on immediate emotional support and connecting students to resources.
  DBT: A structured program that teaches coping skills, emotional regulation, and interpersonal effectiveness.
  Interventions: Behavioral: Psychological First Aid versus Dialectal behavioral Intervention
- Control (Active Comparator): Group A: Begins with PFA followed by DBT. Group B: Begins with DBT followed by PFA.
  Interventions: Behavioral: Psychological First Aid versus Dialectal behavioral Intervention

INTERVENTIONS:
Behavioral: Psychological First Aid versus Dialectal behavioral Intervention — PFA is an immediate, supportive intervention aimed at helping individuals in distress. It focuses on providing emotional support and practical assistance in the aftermath of a crisis.
  Key Components:
  Safety and Comfort: Ensuring that participants feel safe and secure in their environment.
  Active Listening: Engaging in empathetic listening to validate participants' feelings and experiences.
  Assessment of Needs: Identifying immediate needs and concerns, including emotional and practical aspects.
  Information and Resources: Providing clear information about available resources, such as mental health services and coping strategies.
  Encouragement of Social Support: Guiding participants to connect with friends, family, or support groups.

SUMMARY:
his feasibility study aims to compare the effectiveness of Psychological First Aid (PFA) and Dialectical Behavior Therapy (DBT) interventions in reducing suicide risk among undergraduate students. The study employs a crossover randomized controlled trial design, allowing participants to experience both interventions at different times.

DETAILED DESCRIPTION:
Suicide risk among undergraduate students is a pressing mental health concern, exacerbated by academic pressures and social isolation. Psychological First Aid (PFA) is a supportive intervention designed to reduce distress and foster coping in the immediate aftermath of a crisis. Conversely, Dialectical Behavior Therapy (DBT) is a structured, evidence-based therapy that focuses on emotional regulation, interpersonal effectiveness, and distress tolerance. This study explores the feasibility and effectiveness of these two interventions in a university setting.

ELIGIBILITY:
Inclusion Criteria:

Participants in this feasibility study must be undergraduate students aged 18-25 years who are identified as at risk for suicide based on a validated screening tool. They must be currently enrolled in a degree program, able to provide informed consent, and proficient in English.

Exclusion Criteria:

Individuals with severe mental illnesses (e.g., schizophrenia, bipolar disorder), those in acute crisis requiring immediate intervention, current substance abuse issues, significant cognitive impairments, prior experience with DBT or similar therapies within the last year, and physical health conditions that could complicate participation.

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Suicidal Ideation Attributes Scale | 3 months
  It is a brief and reliable tool for assessing the severity of suicidal ideation over the past month, was developed by Van Spijker et al, (2014). It comprises five items that evaluate the frequency of suicidal thoughts, the level of control over these thoughts, proximity to a suicide attempt, the distress caused by the thoughts, and their impact on daily functioning.
The Attitudes Toward Seeking Professional Psychological Help-Short Form | 3 months
  It is a 10-item scale to evaluate attitudes toward seeking psychological help. Responses are rated on a 4-point Likert scale ranging from 0 to 3, with higher scores indicating more favourable attitudes and lower stigma associated with mental illness
Perception of Academic Stress Scale | 3 months
  It was developed by Bedewy, D., & Gabriel, A. (2015), to measure sources of academic stress among university students. PAS IS an 18-item, 5-point Likert-type questionnaire designed, with a higher score indicating higher academic stress.
The Brief Resilience Scale | 3 months
  It is a six-item self-report measure designed to assess resilience by Smith et al. (2008), specifically focusing on an individual's ability to bounce back or recover from stress. Unlike other resilience scales emphasizing resources or traits promoting resilience, the BRS directly evaluates recovery and adaptability following stressful events.
The Self-Compassion Scale | 3 months
  It was developed by Dr. Kristin Neff, is a widely recognized tool designed to measure self-compassion, which encompasses being kind and understanding toward oneself in times of difficulty.

CONTACTS AND LOCATIONS:
Locations (1):
- South Valley Committee, Qina, Egypt